CLINICAL TRIAL: NCT02077933
Title: A Phase Ib Dose-finding Study of BYL719 Plus Everolimus and BYL719 Plus Everolimus Plus Exemestane in Patients With Advanced Solid Tumors, With Dose-expansion Cohorts in Renal Cell Cancer (RCC), Pancreatic Neuroendocrine Tumors (pNETs), and Advanced Breast Cancer (BC) Patients.
Brief Title: Study of Safety and Efficacy of Alpelisib With Everolimus or Alpelisib With Everolimus and Exemestane in Advanced Breast Cancer Patients, Renal Cell Cancer and Pancreatic Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CBYL719Z2102; 2013-004829-86 (EudraCT Number)
Record Dates: First submitted 2014-02-28; First posted 2014-03-04 (Estimated); Last update posted 2020-12-08 (Actual); Status verified 2020-12

CONDITIONS: Neoplasms; Breast Neoplasms; Kidney Neoplasms; Pancreatic Neuroendocine Neoplasms (pNETs)
Keywords: Solid tumors; renal cell carcinoma (RCC); pancreatic neuroendocrine tumors; breast cancer; PI3K inhibitor; BYL719; alpelisib; everolimus; exemestane
MeSH Terms: conditions — Neoplasms; Breast Neoplasms; Kidney Neoplasms; Carcinoma, Renal Cell | interventions — Alpelisib; Everolimus; exemestane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- alpelisib and everolimus (Experimental): alpelisib and everolimus administered once a day
  Interventions: Drug: alpelisib; Drug: everolimus
- alpelisib, everolimus and exemestane (Experimental): alpelisib, everolimus and exemestane administered once a day
  Interventions: Drug: alpelisib; Drug: everolimus; Drug: exemestane
- alpelisib and exemestane (Experimental): alpelisib and exemestane administered once a day
  Interventions: Drug: alpelisib; Drug: exemestane

INTERVENTIONS:
Drug: alpelisib — alpelisib is administered orally once a day on a continuous dosing schedule and dosed on a flat-fixed dose and not adjusted by body weight or body surface area, starting on Day 8 of Cycle 1 in the dose escalation and Day 1 of Cycle 1 in the dose expansion.
  In the doublet dose escalation, the alpelisib starting dose is 300 mg. The alpelisib dose may be escalated or de-escalated, as needed.
  In the triplet dose escalation part, the alpelisib starting dose is one dose level lower of the MTD as determined during the doublet escalation. The alpelisib dose may be escalated or de-escalated, as needed.
  In the doublet dose expansion and triplet dose expansion (patients assigned to alpelisib, everolimus and exemestane), alpelisib is administered at the recommended dose determined in the dose escalation.
  In the triplet dose expansion (patients assigned to alpelisib and exemestane), alpelisib is administered at a dose of 250 mg daily.
Drug: everolimus — everolimus is administered orally once a day on a continuous dosing schedule and dosed on a flat-fixed dose and not adjusted by body weight or body surface area, starting on Day 1 of cycle 1 in both the dose escalation and dose expansion parts.
  In the dose escalation part, the everolimus starting dose is 2,5 mg. In the dose expansion part, everolimus is administered at the recommended dose determined in the dose escalation.
  Arms: alpelisib and everolimus; alpelisib, everolimus and exemestane
Drug: exemestane — exemestane is administered orally once a day on a continuous dose of 25 mg starting on Day 1 of Cycle 1 in both the dose escalation and dose expansion.
  Arms: alpelisib and exemestane; alpelisib, everolimus and exemestane

SUMMARY:
Dose escalation part: to determine the highest dose of alpelisib administered on a daily basis when given in combination with daily everolimus or in combination with daily everolimus and exemestane.

Dose expansion part: To describe safety and tolerability of the alpelisib and everolimus or alpelisib, everolimus and exemestane combinations.

DETAILED DESCRIPTION:
The main purpose of the study was to determine the maximum tolerated dose/recommended dose for expansion (MTD/RDE) of alpelisib in combination with everolimus, and of alpelisib in combination with everolimus and exemestane, and additionally to describe safety, preliminary efficacy and the magnitude of the alpelisib-everolimus interaction. The study was conducted in patients with metastatic and/or recurrent solid tumors including renal cell carcinoma (RCC), pancreatic neuroendocrine tumor (pNET), and advanced solid tumors previously treated with an mTOR inhibitor, to evaluate everolimus and alpelisib, and in postmenopausal females with HR-positive HER2-negative advanced breast cancer to evaluate everolimus, alpelisib and exemestane.

This was a Phase Ib, open-label, multi-center, dose-finding study. The initial dose level of alpelisib was 300 mg every day (qd) and everolimus was initially administered at 2.5 mg qd. The dose-finding study (escalation phase) was followed by an expansion phase where safety and preliminary efficacy of the doublet (alpelisib and everolimus) as well as of the triplet (alpelisib, everolimus and exemestane) were assessed in selected subject populations.

Alpelisib, everolimus and exemestane were administered orally once daily on a continuous dosing schedule and dosed on a flat-fixed dose and not by body weight or body surface area, starting on Day 1 in a 28-day cycle.

In the doublet escalation phase, alpelisib was administered at 300 mg or 250 mg in combination with 2.5 mg everolimus. In the triplet escalation phase, alpelisib was administered at 200 mg in combination with 2.5 mg everolimus and 25 mg exemestane.

In the doublet expansion phase, alpelisib was administered at 250 mg in combination with 2.5 mg everolimus. In the breast cancer expansion phase, alpelisib was administered at 200 mg in combination with 2.5 mg everolimus and 25 mg exemestane or alpelisib was administered at 250 mg in combination with 25 mg exemestane.

No fixed treatment duration was specified. Patients in the study were planned to receive the treatment until disease progression (assessed by Response Evaluation Criteria in Solid Tumors (RECIST v1.1)), unacceptable toxicity, death, or discontinuation from study treatment for any other reason.

ELIGIBILITY:
Inclusion Criteria For entire trial:

* Adult > or = 18 years old
* has signed the Informed Consent Form
* has tumor tissue available for the analysis as described in the protocol
* has an Eastern Cooperative Oncology Group performance status ≤2
* has adequate bone marrow and organ function as defined in the protocol
* is able to swallow and retain oral medication
* has either measurable or non-measurable disease as per RECIST 1.1.

Inclusion Criteria for the BYL719+ Everolimus combination - escalation phase - all above plus has a histologically/cytologically confirmed metastatic and/or recurrent solid tumors for whom no standard therapy exists.

Inclusion Criteria for the BYL719+ Everolimus combination - expansion phase, renal cell carcinoma cohort - all of above first 7 criteria plus has an histologically/cytologically confirmed Renal Cell Cancer as detailed in the protocol

Inclusion Criteria for the BYL719+ Everolimus combination - expansion phase, pancreatic NeuroEndocrine Tumor cohort

- all of above first 7 criteria plus has an histologically/cytologically confirmed pancreatic NeuroEndocrine Tumor as detailed in the protocol

Inclusion Criteria for the BYL719+ Everolimus combination - expansion phase, mTOR inhibitor-pretreated patients' cohort - all of above first 7 criteria plus has a histologically and/or cytologically confirmed solid malignancy as described in the protocol

Inclusion Criteria for the breast cancer cohorts in escalation and expansion phases, - all of above first 7 criteria plus is post-menopausal and has a histologically and/or cytologically confirmed diagnosis of breast cancer as described in the protocol

Specific Inclusion Criteria at the time of cross-over (breast cancer, expansion phase),

- Patient randomized to the alpelisib and exemestane combination who has a radiologically documented progressive disease as detailed in the protocol

Exclusion Criteria:

* Patient has received previous treatment with a PI3K and/or AKT and/or mTOR inhibitor (mTOR inhibitor is allowed in expansion cohorts where patients should have areceived a prior mTOR inhibitor)
* Known intolerance or hypersensitivity to Everolimus or other rapamycin analogs
* Patient with primary central nervous system (CNS) tumor or CNS tumor involvement as detailed in the protocol
* Patient with diabetes mellitus, or documented steroid-induced diabetes mellitus
* Patient has a history of another malignancy within 2 years prior to starting study treatment as described in the protocol
* Patient who has not recovered to grade 1 or better (except alopecia) from related side effects of any prior antineoplastic therapy as detailed in the protocol
* Patient who has had systemic therapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to starting study treatment
* Patient who has received radiotherapy ≤ 4 weeks prior to starting study drugs, with exception of palliative radiotherapy (≤ 2 weeks prior to starting study drugs), who has not recovered from side effects of such therapy to baseline or Grade ≤ 1 and/or from whom ≥ 30% of the bone marrow was irradiated
* Patient who has undergone major surgery ≤ 4 weeks prior to starting study treatment or who has not recovered from side effects of such procedure
* Patient has a clinically significant cardiac disease or impaired cardiac function or any severe and/or uncontrolled medical conditions as detailed in the protocol
* Patient who is currently receiving medication with a known risk of prolonging the QT interval or inducing Torsades de Pointes (TdP) and the treatment cannot either be discontinued or switched to a different medication prior to starting study drug treatment
* Patient who has participated in a prior investigational study within 30 days prior to enrollment as described in the protocol
* Patient who is currently receiving treatment with drugs known to be moderate or strong inhibitors or inducers of isoenzymes CYP34A or CYP2C8 as described in the protocol. Switching to a different medication prior to start of treatment is allowed
* Patient with impaired gastrointestinal (GI) function or GI disease that may significantly alter the absorption of oral alpelisib, everolimus, exemestane
* Patient with known positive serology for human immunodeficiency virus
* Patients who have received live attenuated vaccines within 1 week of start of study drug and during the study as specified in the protocol.
* Pregnant or nursing (lactating) woman as detailed in the protocol.
* Patient who does not apply highly effective contraception during the study and through the duration as defined in the protocol
* Patients in the mTOR inhibitor-pretreated cohorts: all of above first 19 criteria plus have discontinued prior mTOR inhibitor therapy due to non-tolerable toxicity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2014-05-14 (Actual); Primary Completion 2019-04-12 (Actual); Study Completion 2019-04-12 (Actual)

PRIMARY OUTCOMES:
Dose escalation : Incidence of dose Limiting Toxicity (DLTs) | First 35 days of treatment
  To determine the MTD and/or RDE of alpelisib in combination with everolimus, and the MTD and/or RDE of alpelisib in combination with everolimus and exemestane.
  A dose-limiting toxicity (DLT) is an adverse event or abnormal laboratory value assessed as being unrelated to disease, disease progression, inter-current illness, or concomitant medications, and that occurs within the first 35 days of treatment with alpelisib plus everolimus or alpelisib plus everolimus plus exemestane and meets any of the pre-defined criteria.
Dose expansion: Number of patients with adverse events as a measure of safety and tolerability | Screening, every 28 days until 30 days after last dose
  Type, intensity, severity and seriousness of adverse events according to the National Cancer Institute Common Terminology Criteria for Advers Events (NCI CTC AE) v4.03. Dose interruptions, reductions and dose intensity

SECONDARY OUTCOMES:
Dose escalation: Number of patients with adverse events as a measure of safety and tolerability | Screening, every 28 days, until 30 days after last dose
  type, intensity, severity and seriousness of adverse events according to the NCI CTC AE v4.03. Dose interruptions, reductions and dose intensity
Dose escalation : alpelisib, everolimus and exemestane (when applicable) Plasma concentrations | Cycle 1 Day 7, Cycle 1 Day 8, Cycle 1 Day 15, Cycle 1 Day 16, Cycle 1 Day 22, Cycle 2 Day 1, Cycle 2 Day 2, Cycle 2 Day 15, Day 1 of each subsequent cycle
  Plasma concentration time profiles of alpelisib , BZG791, everolimus and exemestane (when applicable). Plasma PK parameters of everolimus, alpelisib, BZG791 and exemestane (when applicable)
Dose escalation : alpelisib, everolimus drug-drug interaction | Cycle 1 Day 7, Cycle 1 Day 8, Cycle 1 Day 15, Cycle 1 Day 16, Cycle 1 Day 22, Cycle 2 Day 1, Cycle 2 Day 2, Cycle 2 Day 15, Day 1 of each subsequent cycle
  Plasma PK parameters of everolimus including AUC ratio (single agent vs. combination)
Dose expansion: Progression free survival (Doublet cohorts) | Baseline, every 8 weeks until first documented disease progression up to 2.5 years.
  Progression-free survival is defined as the time from start date of study treatment until objective tumor progression or death from any cause.
Dose expansion : Duration of Response (Doublet and breast cancer cohorts) | Baseline, every 8 weeks until first documented disease progressionup to 2.5 years.
  Duration of response is defined as the time of first occurrence of Complete Response or Partial Response until the date of the first documented disease progression or death due to the disease.
Dose expansion: Clinical benefit Rate (Doublet and breast cancer cohorts) | Baseline, every 8 weeks until first documented disease progression up to 2.5 years.
  Clinical benefit rate is defined as the proportion of patients with a best overall response of complete response (CR) or partial response (PR) or stable disease (SD) for more than 24 weeks.
Dose expansion: Overall response rate (Doublet and breast cancer cohorts) | Baseline, every 8 weeks until first documented disease progression up to 2.5 years.
  Overall response rate is defined as the proportion of patients with a best overall response of complete response (CR) or partial response (PR), based on RECIST 1.1 criteria and the investigator assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (19):
- United States (2):
  - Highlands Oncology Group, Fayetteville, Arkansas
  - Memorial Sloan Kettering Cancer Center SC - BYL719Z2102, New York, New York
- France (3):
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Villejuif
- Germany (3):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Hanover
- Novartis Investigative Site, Hong Kong, Hong Kong
- Novartis Investigative Site, Budapest, Hungary
- Italy (4):
  - Novartis Investigative Site, Ancona, AN
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Modena, MO
  - Novartis Investigative Site, Verona, VR
- Netherlands (2):
  - Novartis Investigative Site, Amsterdam
  - Novartis Investigative Site, Utrecht
- Spain (2):
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Madrid
- Novartis Investigative Site, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fankhauser M, Bechmann N, Lauseker M, Goncalves J, Favier J, Klink B, William D, Gieldon L, Maurer J, Spottl G, Rank P, Knosel T, Orth M, Ziegler CG, Aristizabal Prada ET, Rubinstein G, Fassnacht M, Spitzweg C, Grossman AB, Pacak K, Beuschlein F, Bornstein SR, Eisenhofer G, Auernhammer CJ, Reincke M, Nolting S. Synergistic Highly Potent Targeted Drug Combinations in Different Pheochromocytoma Models Including Human Tumor Cultures. Endocrinology. 2019 Nov 1;160(11):2600-2617. doi: 10.1210/en.2019-00410. PMID 31322702
- See also: Novartis Clinical Trial Results Database — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=17630